CLINICAL TRIAL: NCT06252870
Title: Randomized Phase 2 Study Testing Two Conditioning Regimen With a Single Prophylaxis of Graft-versus-host Disease by Cyclophosphamide and Methotrexate Post-transplant in Patients Eligible for Matched-donor Allograft Transplantation
Brief Title: Study Testing Two Conditioning Regimen With a Single Prophylaxis of GVHD by Cyclophosphamide and Methotrexate Post-transplant in Patients Eligible for Matched-donor Allograft Transplantation
Acronym: CY-MET-RIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC23_0286
Record Dates: First submitted 2024-01-24; First posted 2024-02-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Graft Versus Host Disease; Hematologic Malignancy
Keywords: Hematopoietic stem cell allograft (Allo-CSH); Methotrexate (MTX); Post-transplant cyclophosphamide (PTCY)
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms | interventions — Methotrexate; fludarabine; Whole-Body Irradiation; Clofarabine; Thiotepa; Busulfan

STUDY DESIGN:
Intervention Model Description: Multicenter, phase 2, non-comparative, randomized, open-label, prospective drug trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (CLO)-BALTIMORE (Experimental): BALTIMORE conditioning regime for LYMPHOID HEMOPATHY CLO-BALTIMORE conditioning regime for MYELOID HEMOPATHY
  Interventions: Drug: Methotrexate; Drug: Post-Transplant Cyclophosphamide; Drug: Fludarabine; Drug: Cycophosphamide; Drug: Anti-Thymoglobulin; Radiation: total body irradiation; Other: hematopoietic stem cells; Other: Graft nuclear cells; Other: Donor Lymphocytes Injection; Drug: Clofarabine
- TBF (Active Comparator): Conditioning regimen for LYMPHOID AND MYELOID HEMOPATHY
  Interventions: Drug: Methotrexate; Drug: Post-Transplant Cyclophosphamide; Drug: Anti-Thymoglobulin; Other: hematopoietic stem cells; Other: Graft nuclear cells; Other: Donor Lymphocytes Injection; Drug: Thiotepa; Drug: Busulfan; Drug: Fludarabine

INTERVENTIONS:
Drug: Methotrexate — 15 mg/m² on Day+1 after graft (=Day0) 10 mg/m² 3 days on Day+4/Day+6/Day+11 after graft (=Day0)
  Other Names: MTX
Drug: Post-Transplant Cyclophosphamide — 50 mg/kg intravenous 2 days on Day+3/Day+5 after graft (=Day0)
  Other Names: CY
Drug: Fludarabine — Conditioning regimen: 30 mg/m² Intravenous 5 days from Day-6 to Day-2 (Day-6/Day-5-/Day-4/Day-3/Day-2 before graft (=Day0)
  Other Names: Fludarabine Baltimore
  Arms: (CLO)-BALTIMORE
Drug: Cycophosphamide — Conditioning regimen: 14.5 mg/kg intravenous 2 days on Day-6/Day-5 before graft (=Day0)
  Arms: (CLO)-BALTIMORE
Drug: Anti-Thymoglobulin — Conditioning regimen: 2.5 mg/kg intravenous on Day-2 before graft (=Day0)
  Other Names: ATG
Radiation: total body irradiation — 2 grays on Day-1 before graft (=Day0)
  Other Names: TBI
  Arms: (CLO)-BALTIMORE
Other: hematopoietic stem cells — High dose of hematopoietic stem cells derived from peripheral blood on transplantation day (=Day0 graft)
  Other Names: HSC
Other: Graft nuclear cells — Graft nuclear cells CD3+ cells if needed after transplantation
Other: Donor Lymphocytes Injection — DLI with CD3+ if relapse after transplantation or in prevention of relapse
  Other Names: DLI
Drug: Clofarabine — Conditioning regimen: 30 mg/m² Intravenous 5 days from Day-6 to Day-2 (Day-6/Day-5-/Day-4/Day-3/Day-2 before graft (=Day0)
  Arms: (CLO)-BALTIMORE
Drug: Thiotepa — Conditioning regimen: 5 mg/kg Intravenous at Day-6 before graft (=Day0)
  Arms: TBF
Drug: Busulfan — Conditioning regimen: 3.2 mg/kg Intravenous 2 days at Day-2 and Day-1 before graft (=Day0)
  Arms: TBF
Drug: Fludarabine — Conditioning regimen: 40 mg/m² intravenous 4 days on Day-5/Day-4/Day-3/Day-2 before graft (=Day0)
  Other Names: Fludarabine TBF
  Arms: TBF

SUMMARY:
Graft-versus-host disease (GVHD) is a major complication of allogeneic hematopoietic stem cell transplantation (allo-CSH).

Recently, in the context of semi-identical (=haploidentical) HLA donors, but also of compatible HLA donors, the use of cyclophosphamide (CY) administered in high doses at early post-transplant (PT) (=PTCY) (Days +3 and +4 or +5) has shown excellent control of acute and chronic GVH, even enabling the discontinuation of other immunosuppressive drugs administered after allo-CSH (ciclosporin, mycophenolate mofetyl (MMF) or Cellcept).

This step has already been taken in the context of allo-CSH with myeloablative conditioning (MAC), which is a minoritary conditioning in adults.

However, in the context of allo-CSH with reduced-intensity conditioning (RIC), which predominates in adults, this strategy seems insufficient to prevent the risk of GVHD.

The idea of reducing the use of immunosuppressants in the context of RIC/HLA-compatible transplants seems, however, still relevant, in order to reduce their adverse effects, improve patients' quality of life and enhance the reconstitution of the post-transplant immune system.

DETAILED DESCRIPTION:
For this reason, the investigators now wish to test the administration of a combination of a high dose of early post-transplant CY (PTCY) and methotrexate (MTX) on days (D) D+1, D+4, D+6, D+11 (doses already performed in MAC transplant prophylaxis), with anti-lymphocyte serum (ALS) with RIC conditioning, without ciclosporin or MMF.

The investigators hypothesize that administration of this PTCY+MTX combination will enable immunosuppressive drugs to be discontinued as early as D+11 post-transplant, compared with the usual average of 3 to 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 and ≤ 70 years old
* Patient with hematologic malignancy
* Indication for HSC allograft with attenuated conditioning
* Pluripotent stem cell (PSC) engraftment
* Availability of a 10/10 familial or non-familial HLA compatible donor
* Consent to the protocol
* ECOG <=2
* Woman of childbearing age with negative pregnancy test and on highly effective contraception during treatment and for a period of 12 months after stopping MTX and CY
* Man of childbearing age with highly effective contraception during treatment and for a period of 6 months after stopping MTX and CY and a period of 12 months after stopping MTX and CY if TBF conditioning regimen arm
* Negative Hepatitis B, C, HIV serologies
* Social security affiliation

Exclusion Criteria:

* History of allograft
* Patient eligible for myeloablative conditioning (MAC)
* Bone marrow transplant
* Other progressive cancerous disease, or antecedent of cancer in the last five years, with the exception of a carcinoma of the skin or a carcinoma in situ of the uterine cole treated and in remission.
* Progressive psychiatric condition
* Pregnant or breastfeeding woman,
* Woman or man of childbearing age with lack of effective contraception
* Serious and uncontrolled concomitant infection
* Cardiac: systolic ejection fraction < 50% by transthoracic ultrasound or by isotopic method (isotope gamma angiography), NYHA II, III or IV heart failure, active rhythmic, valvular or ischemic heart disease or anteriority
* Respiratory with EFR: DLCOc <40% of theoretical
* Renal: creatinine clearance < 50 ml/min (assessment with MDRD method)
* Urological: active urinary tract infection, history of acute urothelial toxicity due to cytotoxic chemotherapy or radiotherapy, known obstruction of urinary flow, pre-existing hemorrhagic cystitis
* Hepatic: transaminases greater than 5 times normal or bilirubin greater than 2 times normal
* Person protected by law (major under guardianship, curatorship or legal protection)
* Vaccination against yellow fever in the last year
* Known or suspected hypersensitivity to rabbit proteins as well as to the active substance and excipients of all investigational and ancillary drugs administered during the study,
* Contraindication to any of the investigational or adjuvant drugs administered during the study
* Patient not speaking French

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2027-10-18 (Estimated); Study Completion 2028-07-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3-4 acute GVHD following allo-CSH for all patients and for each conditioning group (Baltimore and TBF). | Post-transplant through study completion, an average of 1 year
  Estimation of the incidence of grade 3 and 4 acute GVHD following allo-CSH (excluding post-DLI* acute GVHD) according to Mount Sinai criteria.

SECONDARY OUTCOMES:
Incidence of engraftment | Month 1 post-transplant
  Engraftment assessed on hematological reconstitution (number of days of aplasia with PNN <0.5 G/L and platelets < 20 G/L, number of platelet and red cell concentrate transfusions)
Overall survival (OS) | Post-transplant through study completion, an average of 1 year
  survival between day 0 of transplantation and date of death or last follow-up
Disease-free survival (DFS) | Post-transplant through study completion, an average of 1 year
  survival between day 0 of transplantation and date of relapse, death or last follow-up
GVHD and relapse-free survival (GRFS) | Post-transplant through study completion, an average of 1 year
  relapse-free survival without grade 3-4 acute GVHD or chronic GVHD requiring systemic treatment
Incidence of acute GVHD grade 2-4 | Post-transplant through study completion, an average of 1 year
  Acute GVH grade 2-4 according to Mount Sinai criteria
Incidence of chronic GVHD | From month 3 post-transplant through study completion, an average of 1 year
  Chronic GVHD according to NCI criteria
Incidence of corticoresistant acute GVHD | Post-transplant through study completion, an average of 1 year
  Acute corticoresistant GVHD according to the criteria of Mohty et al. defined by :
  * worsening/progression of disease after 3 days of 2mg/kg/day systemic corticosteroid therapy with methylprednisolone (or equivalent),
  * non-improvement of disease after 7 days of 2mg/kg/day systemic corticosteroid therapy with methylprednisolone (or equivalent),
  * disease progression to a new organ after treatment with 1mg/kg/day methylprednisolone (or equivalent) in the case of cutaneous or gastrointestinal GVHD or,
  * recurrence of acute GVHD during or after the corticosteroid reduction phase
Incidence of non-relapse mortality (NRM) | Post-transplant through study completion, an average of 1 year
  any death unrelated to relapse or disease progression
Incidence of relapse | Post-transplant through study completion, an average of 1 year
  any documented disease recurrence
Chimerism | At Month1, Month2, Month3, Month6, Month12 post-transplant
  Total donor or mixed chimerism. Total donor chimerism = result >95% donor CD3+ cells. Mixed chimerism = result >5% and <95% donor CD3+ cells.
Immune reconstitution | At Month3, Month6, Month9, Month12 post-transplant
  T, NK, B lymphocytes and monocytes
Grade 3 and 4 post-transplant adverse events | Post-transplant through study completion, an average of 1 year
  Grade 3 and 4 post-transplant adverse events (dates of occurrence) (NCI CTCAE criteria, version number 5)
Incidence of viral, bacteriological, fungal and parasitic infections | Post-transplant through study completion, an average of 1 year
  Infections: viral (CMV, EBV, BKV, adenovirus), bacteriological, fungal and parasitic

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain THEPOT, MD, Principal Investigator — Angers University Hospital; Marie-Anne COUTURIER, MD, Principal Investigator — University Hospital, Brest
Locations (3):
- France (3):
  - CHU Angers, Angers
  - CHU Brest, Brest
  - CHU Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No